CLINICAL TRIAL: NCT03826576
Title: A Restaurant-based Intervention to Promote Healthy and Allergy Adapted Diet: A Randomized Controlled Trial in Tarragona (Spain)
Brief Title: Healthy Meals: A Restaurant-based Study to Promote Healthy and Allergy Adapted Diet
Acronym: HealthyMeals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Rovira i Virgili (Other)
Collaborators: Diputació de Tarragona (Unknown)
Responsible Party: Principal Investigator, Rosa Sola, Full Professor, MD, PhD, University Rovira i Virgili
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Healthy Meals
Record Dates: First submitted 2019-01-25; First posted 2019-02-01 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Intervention; Food Allergy; Food Preferences; Food Intolerance; Diet Habit; Diet Modification
Keywords: mediterranean diet; Food allergen; restaurant-based intervention
MeSH Terms: conditions — Food Hypersensitivity; Food Preferences; Food Intolerance; Feeding Behavior

STUDY DESIGN:
Intervention Model Description: Parallel randomized controlled trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Intervention group will receive a Multicomponent Intervention.
  Interventions: Behavioral: Multicomponent intervention
- Control Group (No Intervention): Control group will not receive any kind of intervention, only it will receive information about AMED criteria and allergens of food.

INTERVENTIONS:
Behavioral: Multicomponent intervention — The multicomponent intervention will be consist of:
  1. Training of the restaurant staff (waiters and cookers) about Mediterranean and Healthy Diet and food allergens,
  2. Nutritional and food allergen analysis of the menu of the restaurant
  3. Improvement of the menu to follow the Mediterranian diet standards (AMED criteria), the nutritional quality of the menu and the adaptations of the menu for food allergies and food intolerances
  4. Marketing campaign about healthy and food allergen adapted menus in the restaurants
  Arms: Intervention Group

SUMMARY:
This study evaluates the effect of a multicomponent intervention applied to restaurant staff about training and nutritional quality of menu improvement, in order to promote a healthy diet and a better management of allergies and intolerances addressed to each family member satisfying the customers with specific needs (allergies and intolerances of food).

DETAILED DESCRIPTION:
The aim is to test the effect of a multicomponent intervention applied to restaurant staff about training and nutritional quality of menu improvement, in order to promote a healthy diet and a better management of allergies and intolerances addressed to each family member satisfying the customers with specific needs (allergies and intolerances of food).

The study is a 12-month restaurant-based intervention study, randomized, controlled and parallel.

ELIGIBILITY:
The inclusion and exclusion criteria were about restaurants, as a unit of randomization. This study is randomized.

Inclusion Criteria:

* to have signed informed consent by the restaurant owner,
* to have minimum 5 tables of service,
* to offer local or Mediterranean food and recipes on the menu,
* to have the recipes with ingredient and cooking steps details, and
* to share the food products information used in the restaurant with the research team.

Exclusion Criteria:

* To be an ethnic restaurant, fast-food restaurant or a restaurant with a single product like only pizza, sushi, etc
* Lack of one of the inclusion criteria

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2019-02-21 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-12-22 (Actual)

PRIMARY OUTCOMES:
Number of restaurants that accomplish the nine compulsory criteria of the Mediterranean Diet certification (AMED certfication) | 12 months
  Number of restaurants that accomplish the nine compulsory criteria of the Mediterranean Diet certification (AMED certfication). The Mediterranean Diet criteria (AMED Criteria) is a questionnaire based on 9 compulsory criteria, and if the restaurants accomplish this criteria could request the certification of the Mediterranean Diet in their restaurant.
Number of dishes per restaurant that have green colour in Traffic light system | 12 months
  Number of dishes offered in the restaurant with green (good nutritional quality) in the traffic light system, used to measure the nutritional quality.
Number of dishes offered without food allergens, or vegeterian/vegan options | 12 months
  Number of dishes offered without food allergens, or vegeterian/vegan options
Grams of macronutrients in the dishes offered in the restaurants | 12 months
  Reduction of salt, saturated fat and sugar; and increase of fiber in the dishes offered in the restaurants.
  The improvement of nutritional quality of the dishes offered in the restaurant menu through macronutrients assessment.

SECONDARY OUTCOMES:
Number of healthy dishes offered in the restaurants | 12 months
  Number of healthy dishes offered in the restaurants. The healthy dishes considers dishes with traffic light in green in all the macronutrients (sugar, saturated fat, protein, and fiber).
Number of healthy dishes sale in the restaurants | 12 months
  Number of healthy dishes sale in the restaurants. The healthy dishes considers dishes with traffic light in green in all the macronutrients (sugar, saturated fat, protein, and fiber).
Rate of customers with high satisfaction about menu options | 12 months
  Survey of satisfaction
Rate of restaurant staff with high knowledge about healthy and Mediterranean diet, and about food allergens. | 12 months
  Increase the knowledge of waiters and cookers of participant restaurants about healthy and Mediterranean diet, and about food allergens management and options
Annual profits per restaurant in euros | 12 months
  Annual profits per restaurant in euros

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Solà, Prof., Principal Investigator — University Rovira i Virgili
Locations (1):
- Universitat Rovira i Virgili, Reus, Tarragona, Spain

IPD SHARING:
Plan to Share IPD: No